CLINICAL TRIAL: NCT03377491
Title: Pivotal, Randomized, Open-label Study of Tumor Treating Fields (TTFields, 150kHz) Concomitant With Gemcitabine and Nab-paclitaxel for Front-line Treatment of Locally-advanced Pancreatic Adenocarcinoma
Brief Title: Effect of Tumor Treating Fields (TTFields, 150 kHz) as Front-Line Treatment of Locally-advanced Pancreatic Adenocarcinoma Concomitant With Gemcitabine and Nab-paclitaxel (PANOVA-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-27
Record Dates: First submitted 2017-12-06; First posted 2017-12-19 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pancreas Adenocarcinoma
Keywords: Locally Advanced Pancreatic Adenocarcinoma; TTFields; Tumor Treating Fields; Gemcitabine; nab-Paclitaxel; Minimal toxicity; TTF; Novocure
MeSH Terms: interventions — Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- NovoTTF-200T (Experimental): Patients receive TTFields using the NovoTTF-200T System together with gemcitabine and nab-Paclitaxel
  Interventions: Device: NovoTTF-200T; Drug: Gemcitabine; Drug: nab paclitaxel
- Best Standard of Care (Active Comparator): Patients receive best standard of care with gemcitabine and nab-Paclitaxel
  Interventions: Drug: Gemcitabine; Drug: nab paclitaxel

INTERVENTIONS:
Device: NovoTTF-200T — Patients receive continuous TTFields treatment using the NovoTTF-200T device. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the torso. The treatment enables the patient to maintain regular daily routine.
  Other Names: TTFields
  Arms: NovoTTF-200T
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 over 30 minute infusion will be administered immediately after nab-paclitaxel on Days 1, 8 and 15 of each 28-day cycle.
Drug: nab paclitaxel — nab-paclitaxel 125 mg/m^2 administered as an intravenous infusion over 30-40 minutes on Days 1, 8 and 15 of each 28-day cycle.

SUMMARY:
Brief Summary:

The study is a prospective, randomized controlled phase III trial aimed to test the efficacy and safety of Tumor Treating Fields (TTFields) in combination with gemcitabine and nab-paclitaxel, for front line treatment of locally-advanced pancreatic adenocarcinoma.The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE-CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields (TTFields, TTF) has demonstrated significant activity in in vitro and in vivo pancreatic adenocarcinoma pre-clinical models both as a single modality treatment and in combination with chemotherapies. TTFields have been demonstrated to act synergistically with taxanes and have been shown to be additive when combined with other chemotherapies including gemcitabine. In addition, TTFields have shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

In a pilot study, 40 patients with locally advanced or metastatic pancreatic adenocarcinoma received gemcitabine together with TTFields (150 kHz) or gemcitabine and nab-paclitaxel together with TTFields (150 kHz) applied to the abdomen until disease progression. The combination was well tolerated and the only device-related adverse event was contact dermatitis.

In addition, a phase III trial of Optune® (200 kHz) as monotherapy compared to active chemotherapy in recurrent glioblastoma patients showed TTFields to be equivalent to active chemotherapy in extending survival, associated with minimal toxicity, good quality of life, and activity within the brain (14% response rate) (Stupp R., et al., EJC 2012). Finally, a phase III trial of Optune® combined with maintenance temozolomide compared to maintenance temozolomide alone has shown that combined therapy led to a significant improvement in both progression free survival and overall survival in patients with newly diagnosed glioblastoma without the addition of high grade toxicity and without decline in quality of life (Stupp R., et al., JAMA 2017).

DESCRIPTION OF THE TRIAL:

All patients included in this trial are patients with locally advanced pancreatic adenocarcinoma. In addition, all patients must meet all eligibility criteria.

Eligible patients will be randomly assigned to one of two groups:

1. Patients receive gemcitabine and nab-paclitaxel in combination with TTFields using the NovoTTF-200T System.
2. Patients receive gemcitabine and nab-paclitaxel without TTFields.

Patients will be randomized at a 1:1 ratio. Baseline tests will be performed in patients enrolled in both arms. If assigned to the NovoTTF-200T group, the patients will be treated continuously with the device until progression in the abdomen. On both arms, patients who have progression outside the abdomen will switch to a second line treatment according to local practice.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause electrically-charged cellular components of these cells to change their location within the dividing cell, disrupting their normal function and ultimately leading to cell death. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields interfere with the normal orientation of these tiny motors related to other cellular components since they are electrically-charged as well. As a result of these two effects, tumor cell division is slowed, results in cellular death or reverses after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach. Finally, the frequency of TTFields applied to each type of cancer is specific and may not damage normally dividing cells in healthy tissues.

In conclusion, TTFields hold the promise of serving as a brand new treatment for pancreatic adenocarcinoma with very few side effects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Life expectancy of ≥ 3 months
3. Histological/cytological diagnosis of de novo adenocarcinoma of the pancreas
4. Unresectable, locally advanced stage disease according to the following criteria:

   * Head/uncinate process:

     1. Solid tumor contact with SMA>180°
     2. Solid tumor contact with the CA>180°
     3. Solid tumor contact with the first jejunal SMA branch
     4. Unreconstructible SMV/PV due to tumor involvement or occlusion (can be d/t tumor or bland thrombus)
     5. Contact with most proximal draining jejunal branch into SMV
   * Body and tail

     1. Solid tumor contact of >180° with the SMA or CA
     2. Solid tumor contact with the CA and aortic involvement
     3. Unreconstructible SMV/PV due to tumor involvement or occlusion (can be d/t tumor or bland thrombus)
   * No distant metastasis, including non-regional lymph node metastasis
   * No borderline resectable (per Al-Hawary MM, et al., Radiology 201414)
5. ECOG score 0-2
6. Amenable and assigned by the investigator to receive therapy with gemcitabine and nab-paclitaxel
7. Able to operate the NovoTTF-200T System independently or with the help of a caregiver
8. Signed informed consent form for the study protocol

Exclusion Criteria:

1. Prior palliative treatment (e.g. surgery, radiation) to the tumor
2. Cancer requiring anti-tumor treatment within the 5 years before inclusion, excluding treated stage I prostate cancer, in situ cervical or uterus cancer, in situ breast cancer and non-melanomatous skin cancer.
3. Serious co-morbidities:

   1. Clinically significant (as determined by the investigator) hematological, hepatic and renal dysfunction, defined as: Neutrophil count < 1.5 x 10^9/L and platelet count < 100 x 10^9/L; bilirubin > 1.5 x Upper Limit of Normal (ULN); AST and/or ALT > 2.5 x ULN; and serum creatinine > 1.5 x ULN.
   2. History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary activity results in fatigue, palpitation or dyspnea).
   3. History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the trial.
   4. History of cerebrovascular accident (CVA) within 6 months prior to randomization or that is not stable.
   5. Active infection or serious underlying medical condition that would impair the ability of the patient to receive protocol therapy.
   6. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent.
4. Concurrent anti-tumor therapy beyond gemcitabine and nab-paclitaxel
5. Implantable electronic medical devices in the torso, such as pacemakers
6. Known severe hypersensitivities to medical adhesives or hydrogel, or to one of the chemotherapies used in this trial.
7. Pregnancy or breast-feeding (female patients with reproductive potential and their partners must accept to use effective contraception throughout the entire study period and for 3 months after the end of treatment). All patients who are capable of becoming pregnant must take a pregnancy test which is negative within 72 hours before beginning treatment. The definition of effective contraception is left up to the decision of the investigator.
8. Unable to follow the protocol for medical, psychological, familial, geographic or other reasons.
9. Admitted to an institution by administrative or court order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (199):
- United States (74):
  - Grandview Medical Center, Cancer Center, Birmingham, Alabama
  - Infirmary Cancer Care, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology Associates, PC- HOPE - US Oncology Research, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - Providence Medical Foundation, Fullerton, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Dignity Health - Mercy Cancer Centers, Sacramento, California
  - Sutter Cancer Center Sacramento, Sacramento, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Adventist Health St. Helena - Martin-O'Neil Cancer Center (MOCC), St. Helena, California
  - Associated Neurologists of Southern Connecticut, P.C., Milford, Connecticut
  - Boca Raton Regional Hospital, Lynn Cancer Institute, Boca Raton, Florida
  - Cancer Specialist of North Florida, Fleming Island, Florida
  - Florida Cancer Specialists & Research Institute - Colonial Office, Fort Myers, Florida
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Neuro Oncology, Orlando, Florida
  - BRCR Medical Center INC, Plantation, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Illinois Cancer Specialist - US Oncology Research, Arlington Heights, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Cancer Center, Fairway, Kansas
  - Cotton O'Neil Cancer Center (Stormont-Vail Cancer Center), Topeka, Kansas
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Central Maine Medical Center, Clinical Research Department, Lewiston, Maine
  - University of Maryland Comprehensive Cancer Center, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A - US Oncology Research, Columbia, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, PC, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - MidAmerica Division, Kansas City, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Renown Regional Medical Center & Renown Institute for Cancer, Reno, Nevada
  - Astera Cancer Care, East Brunswick, New Jersey
  - Kaleida Health, Buffalo, New York
  - Bassett Medical Center, Cooperstown, New York
  - New York Hospital Queens, Flushing, New York
  - NYU Langone Arena Oncology, Lake Success, New York
  - White Plains Hospital - Center for Cancer Care, White Plains, New York
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Gabrail Cancer Research Center, Canton, Ohio
  - Toledo Clinic Cancer Centers, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center - US Oncology Research, Eugene, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Vita Medical Associates, P.C., Fountain Hill, Pennsylvania
  - UT/Erlanger Oncology & Hematology, Chattanooga, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Beaumont Mamie McFaddin Ward Cancer Center - US Oncology Research, Beaumont, Texas
  - Texas Oncology - Bedford - US Oncology Reasearch, Bedford, Texas
  - Methodist Regional Cancer Center, Dallas, Texas
  - Texas Oncology - Baylor - US Oncology Research, Dallas, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Gateway - US Oncology Research, El Paso, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Baylor Scott and White Medical Center, Temple, Texas
  - Texas Oncology - Tyler - US Oncology Research, Tyler, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care - US Oncology Research, Roanoke, Virginia
  - Vista Oncology Inc PS, Olympia, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia
- Australia (5):
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
  - Monash Medical Centre, Clayton
  - Sydney Adventist Hospital, Wahroonga
  - Westmead Hosptial, Westmead
- Austria (4):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Wörthersee
  - Medical University Graz, Graz
  - Univ. Klinik für Innere Medizin III der PMU, Salzburg
  - Landes-Krankenhaus Steyr, Steyr
- Belgium (3):
  - Faculté de Médecine Campus Erasme, Anderlecht
  - UZ Leuven, Leuven
  - Clinique Universutaire Saint Luc - Institut Roi Albert II, Woluwe-Saint-Lambert
- Brazil (12):
  - Centro de Pesquisa Clínica e Ensino Florianópolis LTDA, Florianópolis
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - IRPCc - Instituto Ribeirãopretano de Combate ao Câncer, Ribeirão Preto
  - Oncoclinicas Group Botafogo, Rio de Janeiro
  - Instituto D'Or de Pesquisa e Ensino - Rio De Janeiro, Rio de Janeiro
  - Groupo Clinicas Oncologicas Integradas (COI) - Barra da Tijuca, Rio de Janeiro
  - Instituto D´Or de Pesquisa e Ensino - Hospital São Rafael, São Marcos
  - Núcleo de Pesquisa Clínica da Rede São Camilo, São Paulo
  - Clínica OncoStar - REDE D´OR, São Paulo
- Canada (3):
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de I'Universitaire de de Montreal (CHUM), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
- China (18):
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Linyi Cancer Hospital, Linyi, Shandong
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People'S Hospital, Beijing
  - The first hospital of Jilin University, Changchun
  - Guangdong provincial people's hospital, Guangzhou
  - Jilin Guowen Hospital, Jilin
  - Shanghai Changhai Hospital, Shanghai
  - Shanxi Provincial Cancer Hospital, Shanxi
  - Xingtai People's Hospital, Xingtai
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Provincial Peoples Hospital, Zhengzhou
- University Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (5):
  - Masaryk Institute of Oncology, Brno-střed
  - Nemocnice Nový Jičín, Nový Jičín
  - University Hospital Olomouc, Olomouc
  - General University Hospital in Prague, Prague
  - Nemocnice Na Bulovce, Prague
- France (8):
  - Hopital haut-Léveque CHU Bordeaux - Service d'Hépato- Gastroentérologie et d'Oncologie digestive, Pessac, Bordeaux
  - Centre Hospitalier de Bretagne Sud /Site du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Service d'Oncologie médicale du Pr. Andre, Hôpital Saint-Antoine, Paris
  - Hôpital Privé des Côtes d'Armor, Plérin
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Centre de Lutte Contre le Cancer (CLCC) - Centre Paul Strauss, Strasbourg
  - Clinique Sainte Anne - Groupe Hospitalier Saint-Vincent, Strasbourg Oncologie Libérale, Strasbourg
- Germany (7):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Medizinische Hochschule Hannover, Klinik fur Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - VK und K Studien GbR Landshut-Achdorf, Landshut
  - Bonifatius Hospital Hematology and Oncology, Lingen
  - Carl-von-Basedow-klinikum Saalekrei, Merseburg
  - Klinikum München Bogenhausen, Klinik für Gastroenterologie und Gastroenterologische Onkologie, München
  - Universitätsklinikum Ulm, Ulm
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (5):
  - National Institute of Oncology, Budapest
  - Bekes County Hospital, Gyula
  - Bacs-Kiskun County Hospital, Kecskemét
  - Tolna County Hospital, Szekszárd
  - Jasz-Nagykun-Szolnok County Hospital, Szolnok
- Israel (5):
  - Rambam Health Care Campus, Oncology Institute, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Pancreatic Cancer Center - SPCC, Ramat Gan
  - Sourasky Medical Center, Oncology Department, Tel Aviv
- Italy (5):
  - A.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Università Campus Bio-Medico di Rome, Roma
  - Ospedale San Giovanni Calibita Fatebenefratelli Isola Tiberina, Roma
  - A.O.U Città della Salute e della Scienza di Torino, Torino
- Mexico (14):
  - Mediadvance Clinical, Chihuahua City, Chih.
  - Accelerium S de RL de C.V., Monterrey, Nuevo León
  - Centro de Estudios de Alta Especialidad de Sinaloa, ubicado, Mazatlán, Sinaloa
  - Centro de Investigación Médica Aguascalientes (CIMA),, Aguascalientes
  - Clinstile S.A. de C.V.,, Cuauhtémoc
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli
  - Hospitales Star Medica - Luna Parc, Estado de México
  - Universidad Autonoma de Nuevo Leon - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - Oncocenter - Puebla, Puebla City
  - Hospital Angeles San Luis, San Luis Potosí City
  - Centro Potosino de Investigación Médica SC,, San Luis Potosí City
  - Centro Hemato-Oncologico Privado CHOP, Toluca
  - Phylasis Clinicas Research S.de R.L. de C.V. (PCR)-Toluca, Toluca
  - FAICIC Clinical Research, Veracruz
- Poland (5):
  - Oncology Clinic Clinical Hospital of Przemienienia Pańskiego UM in Poznaniu, Poznan
  - Centrum Medyczne MrukMed, Rzeszów
  - Oncology and Radiotherapy Clinic, Oncology Center - Institute, Warsaw
  - Oncology and Radiotherapy Clinic University Clinical Center Non-Invasive Medicine Center, Warsaw
  - Jan Mikulicz-Radecki University Teaching Hospital, Wroclaw
- South Korea (13):
  - Dong-A University Hospital, Seogu, Busan
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Keimyung University, Dongsan hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (9):
  - Instituto Oncòlogico Dr. Rosell, Barcelona
  - Vall d´Hebron University Hospital, Barcelona
  - Hospital General Universitario de Elche, Elche
  - HM Hospitales - Centro Integral Oncologico Clara Campal - CIOCC, Madrid
  - Hospital Universitario Ramon Y Cajal Carretera de Colmenar Viejo, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Clinica Universiatria de Navarra, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Instituto Valenciano de Oncología IVO, Valencia
- Switzerland (2):
  - Hôpital Fribourgeois/Freiburger Spital, Fribourg
  - KS Winterthur, Winterthur

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Giladi M, Schneiderman RS, Porat Y, Munster M, Itzhaki A, Mordechovich D, Cahal S, Kirson ED, Weinberg U, Palti Y. Mitotic disruption and reduced clonogenicity of pancreatic cancer cells in vitro and in vivo by tumor treating fields. Pancreatology. 2014 Jan-Feb;14(1):54-63. doi: 10.1016/j.pan.2013.11.009. Epub 2013 Dec 4. PMID 24555979
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Derived] Babiker HM, Picozzi V, Chandana SR, Melichar B, Kasi A, Gang J, Gallego J, Bullock A, Chunyi H, Wyrwicz L, Hitre E, Osipov A, de la Fouchardiere C, Ales I, Dragovich T, Lee W, Feeney K, Philip P, Ueno M, Van Cutsem E, Seufferlein T, Macarulla T; PANOVA-3 Study Investigators. Tumor Treating Fields With Gemcitabine and Nab-Paclitaxel for Locally Advanced Pancreatic Adenocarcinoma: Randomized, Open-Label, Pivotal Phase III PANOVA-3 Study. J Clin Oncol. 2025 Jul 20;43(21):2350-2360. doi: 10.1200/JCO-25-00746. Epub 2025 May 31. PMID 40448572

RESULTS

PARTICIPANT FLOW:
Groups:
- TTFields + Standard of Care: TTFields were to be delivered until local disease progression. Standard of care treatment was administered until disease progression or intolerable toxicity (Nab-paclitaxel 125 mg/m2 and Gemcitabine 1000 mg/m2 on Days 1, 8, 15 of each 28-day cycle).
- Standard of Care: Standard of care treatment was administered until disease progression or intolerable toxicity (Nab-paclitaxel 125 mg/m2 and Gemcitabine 1000 mg/m2 on Days 1, 8, 15 of each 28-day cycle).
Period: Overall Study
Arm/Group | TTFields + Standard of Care | Standard of Care
Started | 285 | 286
Completed (Participants alive at study end are included under 'Study Closure.') | 0 | 0
Not Completed | 285 | 286
Not completed — Death | 193 | 211
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 42 | 26
Not completed — Study closure | 40 | 37
Not completed — Other | 8 | 9

BASELINE CHARACTERISTICS:
Population: There may be more than 1 lesion present in a participant
Units Other Than Participants: Lesions
Groups:
- Total: Total of all reporting groups
Arm/Group | TTFields + Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 285 | 286 | 571
Number analyzed (Lesions) | 310 | 309 | 619
Age, Continuous [Median (Full Range); unit: Years] | 67 [31 to 90] | 67.5 [40 to 88] | 67 [31 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 161 | 299
  Male | 147 | 125 | 272
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 4 | 13
  Asian | 44 | 44 | 88
  Black or African American | 16 | 14 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 202 | 204 | 406
  Other | 3 | 5 | 8
  Not Reported | 11 | 15 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 123 | 125 | 248
  Eastern Europe | 43 | 42 | 85
  Western Europe and Israel | 62 | 61 | 123
  Rest of World | 57 | 58 | 115
ECOG Performance Status [Count of Participants; unit: Participants] — Population: Measure Description: Participants level of functional ability and the extent of disease affect of their daily life were assessed. A score of 0 indicates a better health condition, and a score of 2 indicates a worse health condition.
  Participants
    0 | 109 | 111 | 220
    1 | 166 | 163 | 329
    2 | 10 | 12 | 22
BMI Group [Count of Participants; unit: Participants]
  < 25 kg/m2 | 166 | 174 | 340
  ≥ 25 kg/m2 | 117 | 108 | 225
  Missing BMI | 2 | 4 | 6
CA19.9 [Count of Participants; unit: Participants]
  Low (≤37 U/mL) | 48 | 44 | 92
  Moderate (38-1,000 U/mL) | 140 | 152 | 292
  High (>1,000 U/mL) | 88 | 79 | 167
  Untested | 9 | 11 | 20
Target Lesion Site [Number; unit: Lesions]
  Head of Pancreas | 164 | 160 | 324
  Body of Pancreas | 82 | 81 | 163
  Tail of Pancreas | 9 | 19 | 28
  Other: Multiple regions in pancreas | 26 | 22 | 48
  Other: Extra-pancreatic | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Overall survival of subjects treated with TTFields concomitant with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer subjects, compared to overall survival of subjects treated with chemotherapy alone, measured as the period between the time of randomization and the time of death.
Time Frame: From randomization until death from any cause or last known alive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
Months | 16.20 [15.01 to 17.97] | 14.16 [12.81 to 15.44]
Statistical Analysis 1: Comparison: TTFields + Standard of Care vs Standard of Care; Test type: Superiority; p = 0.039, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.68 to 0.99]

2. Secondary Outcome: Progression-free Survival of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Progression-free survival of subjects treated with TTFields concomitant with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer subjects, compared to the progression-free survival of subjects treated with chemotherapy alone, measured from the time of randomization and based on CT scans collected on the study, using the revised RECIST V1.1 Criteria.
  Progression is defined using the RECIST 1.1 criteria: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, in addition the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, progression was defined as unequivocal progression (an overall level of substantial worsening in non-target disease) of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: From randomization until radiologic disease progression per RECIST v1.1 or death, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
Months | 10.61 [9.20 to 12.19] | 9.33 [7.59 to 11.07]
Statistical Analysis 1: Comparison: TTFields + Standard of Care vs Standard of Care; Test type: Superiority; p = 0.137, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.68 to 1.05]

3. Secondary Outcome: Local Progression-free Survival of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Local progression-free survival of subjects treated with TTFields concomitant with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer subjects, compared to the local progression-free survival of subjects treated with chemotherapy alone, measured from the time of randomization and based on CT scans collected on the study, using the revised RECIST V1.1 Criteria.
  Local progression is defined per RECIST 1.1 in the absence of distant metastasis: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, in addition the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, progression was defined as unequivocal progression (an overall level of substantial worsening) of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: From randomization until local disease progression per RECIST v1.1 (in the absence of distant metastasis) or death, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
Months | 12.45 [10.68 to 14.52] | 10.41 [9.13 to 11.79]
Statistical Analysis 1: Comparison: TTFields + Standard of Care vs Standard of Care; Test type: Superiority; p = 0.151, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.06]

4. Secondary Outcome: Objective Response Rate of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Objective Response Rate (ORR) was assessed per RECIST v1.1. Complete Response (CR): disappearance of all target and non-target lesions and reduction of pathological lymph nodes to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions from baseline without new lesions or progression of non-target lesions. ORR is defined as the percentage of participants whose best overall response was CR or PR.
Time Frame: From randomization until radiologic disease progression per RECIST v1.1 or end of tumor assessment follow-up.
Population: Per SAP, subjects without evaluable post-baseline tumor assessments (unevaluable/missing follow-up data) were excluded. Only subjects with ORR information per RECIST v1.1 were included, which explains why the analyzed N (244 and 243) is different than the ITT population (285 vs 286).
Measure: Count of Participants; unit: Participants
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 244 | 243
Participants | 88 | 73
Statistical Analysis 1: Comparison: TTFields + Standard of Care vs Standard of Care; Test type: Superiority; p = 0.094, t-test, 1 sided

5. Secondary Outcome: One-year Survival Rate of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: One-year survival rate of subjects treated with TTFields concomitant with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer subjects, compared to the 1-year survival rate of subjects treated with chemotherapy alone.
Time Frame: From randomization through 12 months after randomization.
Population: The 1-year OS rate is a Kaplan-Meier (KM) estimate of survival at 12 months in the ITT population. As a time-to-event estimate incorporating censoring, the percentage may not correspond exactly to a simple whole-number count of participants. KM estimate represents risk-adjusted survival probability.
Measure: Number (95% Confidence Interval); unit: percentage of subjects alive at 1 year
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
percentage of subjects alive at 1 year | 68.1 [62.0 to 73.5] | 60.2 [54.2 to 65.7]
Statistical Analysis 1: Comparison: TTFields + Standard of Care vs Standard of Care; Test type: Superiority; p = 0.029, t-test, 1 sided

6. Secondary Outcome: Quality of Life of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Quality of life deterioration-free survival (DFS) was assessed using the EORTC QLQ-C30 and pancreatic cancer-specific QLQ-PAN26 questionnaires. Higher scores on functional and global health status scales indicate better functioning, whereas higher symptom scores indicate worse symptoms.
  DFS was defined as the time from randomization to the first ≥10-point deterioration from baseline without a subsequent ≥10-point improvement, or death. DFS was evaluated separately for each QoL domain included in the analysis.
Time Frame: From randomization until the first ≥10-point deterioration without subsequent improvement, or death, assessed for the duration of study follow-up.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
Months
  Global health status / Quality of Life | 7.1 [5.7 to 9.4] | 5.7 [4.1 to 7.4]
  Pain (EORTC QLQ-C30) | 10.1 [8.0 to 11.6] | 7.4 [5.9 to 9.0]
  Pancreatic pain (EORTC QLQ-PAN26) | 14.7 [12.0 to 16.5] | 10.2 [8.8 to 12.2]
  Digestive problems (EORTC QLQ-PAN26) | 8.3 [6.1 to 11.2] | 5.7 [4.4 to 7.4]

7. Secondary Outcome: Pain-free Survival of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Pain-free survival was measured as the duration between the time of randomization until a greater than or equal to twenty-point increase from baseline in a patient self-reported visual analogue scale (VAS) was recorded or death, whichever occurred first.
Time Frame: From randomization until a ≥20-point increase from baseline in pain on the patient-reported visual analogue scale (0-100) or death, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
Months | 15.18 [10.28 to 22.77] | 9.13 [7.43 to 12.68]

8. Secondary Outcome: Puncture-free Survival of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Puncture-free survival of subjects treated with TTFields concomitant with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer subjects, compared to puncture-free survival of subjects treated with chemotherapy alone, measured as the duration between randomization until the first need for paracentesis or death, whichever occurs first.
Time Frame: From randomization until the first paracentesis or death, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
months | 22.8 [15.5 to NA] — NA indicates that the upper limit of the 95% confidence interval could not be estimated due to an insufficient number of events beyond the median. | 16.6 [13.1 to NA] — NA indicates that the upper limit of the 95% confidence interval could not be estimated due to an insufficient number of events beyond the median.
Statistical Analysis 1: Comparison: TTFields + Standard of Care vs Standard of Care; Test type: Superiority; p = 0.128, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.57 to 1.08]

9. Secondary Outcome: Resectability Rate of Subjects Treated With TTFields Concomitant With Gemcitabine and Nab-paclitaxel vs Chemotherapy Alone
Description: Resectability rate defined as the number and percentage of patients whose tumors were deemed resectable and who underwent surgery.
Time Frame: From randomization through the end of study follow-up. Surgical resections were captured throughout study follow-up, up to approximately 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | TTFields + Standard of Care | Standard of Care
Number analyzed (Participants) | 285 | 286
Participants | 20 [4.3 to 10.6] | 29 [6.9 to 14.2]
Statistical Analysis 1: Comparison: TTFields + Standard of Care vs Standard of Care; Test type: Superiority; p = 0.9311, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization until last study follow up visit and for 30 days following treatment termination, estimated 4 years
Description: AEs were reported for the safety population, defined as subjects who received any amount of study intervention. The descriptions and grading scales found in the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 are utilized for assessing severity of adverse events in the study. However, the CTCAE does not include a scale that properly describes the skin toxicity associated with the NovoTTF-200T system and a modified grading for TTFields-related skin adverse events was used.
Groups:
- TTFields + Standard of Care: TTFields were to be delivered for at least 18 hours per day on a monthly average until local disease progression. Standard of care treatment was administered until disease progression or intolerable toxicity (Nab-paclitaxel 125 mg/m2 and Gemcitabine 1000 mg/m2 on Days 1, 8, 15 of each 28-day cycle).
Arm/Group | TTFields + Standard of Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 199/274 | 223/273
Serious Adverse Events (participants affected / at risk) | 147/274 | 131/273
Other Adverse Events (participants affected / at risk) | 267/274 | 268/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TTFields + Standard of Care (N=274) | Standard of Care (N=273)
Anaemia (Blood and lymphatic system disorders) | 3 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 4 | 6
Neutropenia (Blood and lymphatic system disorders) | 5 | 2
Jaundice (Blood and lymphatic system disorders) | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 4 | 3
Cardiac failure (Cardiac disorders) | 6 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3
Pericardial effusion (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 7
Colitis (Gastrointestinal disorders) | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 7
Abdominal Pain (Gastrointestinal disorders) | 6 | 2
Duodenal obstruction (Gastrointestinal disorders) | 6 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3
Obstruction gastric (Gastrointestinal disorders) | 2 | 4
Ascites (Gastrointestinal disorders) | 4 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 4
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Duodenal stenosis (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 5
Fatigue (General disorders) | 4 | 3
General physical health deterioration (General disorders) | 1 | 4
Generalized edema (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Edema (General disorders) | 1 | 0
Peripheral edema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 16 | 10
Bile duct obstruction (Hepatobiliary disorders) | 15 | 9
Cholecystitis (Hepatobiliary disorders) | 5 | 5
Bile duct stenosis (Hepatobiliary disorders) | 2 | 2
Gallbladder rupture (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Perforation bile duct (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Sepsis (Infections and infestations) | 19 | 26
Pneumonia (Infections and infestations) | 14 | 9
Infection (Infections and infestations) | 8 | 7
COVID-19 (Infections and infestations) | 5 | 4
Urinary tract infection (Infections and infestations) | 3 | 6
Skin infection (Infections and infestations) | 3 | 4
Bacteraemia (Infections and infestations) | 4 | 2
Abscess (Infections and infestations) | 1 | 4
Biliary tract infection (Infections and infestations) | 4 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 0 | 2
Peritonitis (Infections and infestations) | 2 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Fournier's gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatobiliary infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 2 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Pancreatogenous diabetes (Metabolism and nutrition disorders) | 1 | 0
Starvation ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Device occlusion (Product Issues) | 7 | 1
Stent malfunction (Product Issues) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Completed suicide (Psychiatric disorders) | 0 | 1
Eating disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 6
Renal failure (Renal and urinary disorders) | 1 | 4
Nephritic syndrome (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TTFields + Standard of Care (N=274) | Standard of Care (N=273)
Neutropenia (Blood and lymphatic system disorders) | 171 | 180
Anemia (Blood and lymphatic system disorders) | 161 | 155
Thrombocytopenia (Blood and lymphatic system disorders) | 122 | 132
Leukopenia (Blood and lymphatic system disorders) | 85 | 98
Lymphopenia (Blood and lymphatic system disorders) | 22 | 27
Arrhythmia (Cardiac disorders) | 14 | 14
Diarrhea (Gastrointestinal disorders) | 119 | 123
Nausea (Gastrointestinal disorders) | 107 | 121
Vomiting (Gastrointestinal disorders) | 80 | 77
Abdominal Pain (Gastrointestinal disorders) | 69 | 81
Constipation (Gastrointestinal disorders) | 63 | 57
Abdominal distension (Gastrointestinal disorders) | 25 | 28
Mouth ulceration (Gastrointestinal disorders) | 22 | 28
Dyspepsia (Gastrointestinal disorders) | 20 | 23
Ascites (Gastrointestinal disorders) | 21 | 19
Dry mouth (Gastrointestinal disorders) | 18 | 14
Fatigue (General disorders) | 164 | 148
Peripheral edema (General disorders) | 107 | 99
Pyrexia (General disorders) | 73 | 60
Pain (General disorders) | 39 | 27
Hyperbilirubinemia (Hepatobiliary disorders) | 24 | 14
COVID-19 (Infections and infestations) | 38 | 32
Respiratory tract infection (Infections and infestations) | 32 | 27
Urinary tract infection (Infections and infestations) | 29 | 22
Infection (Infections and infestations) | 33 | 22
Pneumonia (Infections and infestations) | 19 | 12
Skin infection (Infections and infestations) | 16 | 13
Fall (Injury, poisoning and procedural complications) | 19 | 15
Hepatic enzyme increased (Investigations) | 75 | 72
Blood lactate dehydrogenase increased (Investigations) | 13 | 17
Blood creatinine increased (Investigations) | 11 | 18
Anorexia (Metabolism and nutrition disorders) | 93 | 101
Hypokalemia (Metabolism and nutrition disorders) | 63 | 70
Hypoalbuminemia (Metabolism and nutrition disorders) | 43 | 26
Hyperglycemia (Metabolism and nutrition disorders) | 27 | 29
Hyponatremia (Metabolism and nutrition disorders) | 27 | 23
Dehydration (Metabolism and nutrition disorders) | 21 | 20
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 | 25
Hypercalcemia (Metabolism and nutrition disorders) | 19 | 15
Hypoproteinemia (Metabolism and nutrition disorders) | 17 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 70 | 79
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 | 15
Neuropathy peripheral (Nervous system disorders) | 112 | 81
Taste disorder (Nervous system disorders) | 38 | 35
Dizziness (Nervous system disorders) | 37 | 28
Headache (Nervous system disorders) | 20 | 19
Hypoaesthesia (Nervous system disorders) | 21 | 12
Paraesthesia (Nervous system disorders) | 16 | 12
Sleep disorder (Psychiatric disorders) | 38 | 26
Depression (Psychiatric disorders) | 24 | 10
Anxiety (Psychiatric disorders) | 14 | 19
Micturition disorder (Renal and urinary disorders) | 15 | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 39 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 32
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 71 | 86
Rash (Skin and subcutaneous tissue disorders) | 71 | 23
Dermatitis (Skin and subcutaneous tissue disorders) | 82 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 61 | 23
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 49 | 27
Erythema (Skin and subcutaneous tissue disorders) | 36 | 9
Nail disorder (Skin and subcutaneous tissue disorders) | 15 | 16
Skin reaction (Skin and subcutaneous tissue disorders) | 20 | 9
Hypertension (Vascular disorders) | 19 | 27
Hypotension (Vascular disorders) | 28 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines. If patentable information is discovered, additional 60 days are required for review.

DOCUMENTS (2):
  • Study Protocol (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT03377491/Prot_002.pdf
  • Statistical Analysis Plan (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03377491/SAP_003.pdf